CLINICAL TRIAL: NCT01041989
Title: Finnish Geriatric Intervention Study to Prevent Cognitive Impairment and Disability
Acronym: FINGER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Finnish Institute for Health and Welfare (Other Government)
Collaborators: Academy of Finland (Other); University of Helsinki (Other); University of Eastern Finland (Other); University of Oulu (Other); Kuopio Research Institute of Exercise Medicine (Other); Western University, Canada (Other); Karolinska Institutet (Other); Umeå University (Other)
Responsible Party: Principal Investigator, Miia Kivipelto, Professor, Finnish Institute for Health and Welfare
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: THL/TUET 122/2009
Record Dates: First submitted 2010-01-04; First posted 2010-01-05 (Estimated); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Cognitive Impairment; Dementia
Keywords: dementia; cognitive impairment; disability; intervention; elderly; lifestyle counseling
MeSH Terms: conditions — Cognitive Dysfunction; Dementia | interventions — Exercise; Cognitive Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard health counseling at baseline (No Intervention)
- Lifestyle counseling (Experimental): Multi-domain lifestyle counseling including nutritional guidance, increased physical activity, cognitive training, increased social activity and intensive monitoring of vascular and metabolic risk factors.
  Interventions: Behavioral: Nutritional guidance; Behavioral: Exercise; Behavioral: Cognitive training; Other: Reduction of vascular risk factors

INTERVENTIONS:
Behavioral: Nutritional guidance — Individual counseling sessions and group meetings will be organized.
  Arms: Lifestyle counseling
Behavioral: Exercise — Guided muscle strength training and aerobic exercise.
  Arms: Lifestyle counseling
Behavioral: Cognitive training — Cognitive training will be implemented through 8 group sessions lead by a psychologist and a computer-based cognitive training program available to participants via the internet.
  Arms: Lifestyle counseling
Other: Reduction of vascular risk factors — Monitoring and maintenance of metabolic and vascular risk factors
  Arms: Lifestyle counseling

SUMMARY:
This multi-center (6 sites: Helsinki, Kuopio, Oulu, Seinäjoki, Turku, Vantaa) intervention study aims to prevent cognitive impairment, dementia and disability in 60-77 year old persons at an increased dementia risk. The 2-year multi-domain life-style intervention includes nutritional guidance, exercise, cognitive training, increased social activity, and intensive monitoring and management of metabolic and vascular risk factors. The primary outcome is cognitive impairment measured by a sensitive Neuropsychological Test Battery (NTB), and Stroop and Trail Making tests to capture early cognitive impairment typical for both Alzheimer's disease and vascular dementia. We hypothesize that the multi-domain intervention will reduce cognitive impairment in the study group compared to the control group during the initial 2-year intervention period and reduce dementia incidence after the extended follow-up (until at least 300 participants have developed dementia).

ELIGIBILITY:
Inclusion Criteria:

* aged 60-77 years
* dementia Risk Score 6 points or more
* fulfillment of at least one of the following CERAD criteria: i) MMSE: 20-26 points ii) word list memory task (3x10 words): 19 words or less iii) delayed recall: 75% or less

Exclusion Criteria:

* malignant diseases
* dementia
* substantial cognitive decline
* major depression
* symptomatic cardiovascular disease
* revascularisation within 1 year
* severe loss of vision, hearing or communicative ability
* other conditions inhibiting from safe engagement in the prescribed intervention as judged by the study physician
* other conditions preventing from cooperation as judged by the study physician

Ages: 60 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2009-09; Primary Completion 2013-12 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Cognitive impairment assessed with a Neuropsychological Test Battery, and Stroop and Trail Making tests. | 2 years

SECONDARY OUTCOMES:
Depressive symptoms will be assessed using the Zung depression scale. | 2 years
Disability will be assessed using the ADCS-ADL scale | 2 years
Quality of Life will be assessed using the RAND-36 and 15D questionnaires. | 2 years
Utilization of health resources will be assessed using questionnaire and register data. | 2 years
Vascular and metabolic risk factors will be assessed with blood pressure and anthropometric measurements, and laboratory analyses of metabolic biomarkers. | 2 years
Vascular and metabolic morbidity and mortality will be assessed through questionnaire and register data. | 2 years
Changes in dietary biomarker levels will be assessed through laboratory testing. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Miia Kivipelto, professor, Principal Investigator — Finnish Institute for Health and Welfare; Tiina K Laatikainen, professor, Study Director — Finnish Institute for Health and Welfare; Hilkka S Soininen, professor, Study Director — University of Eastern Finland; Jaakko Tuomilehto, professor, Study Director — University of Helsinki; Timo E Strandberg, professor, Study Director — University of Oulu; Raimo Sulkava, professor, Study Director — University of Eastern Finland; Rainer Rauramaa, professor, Study Director — Kuopio Research Institute of Exercise Medicine; Antti Jula, research prof, Study Director — Finnish Institute for Health and Welfare; Markku Peltonen, research professor, Study Director — Finnish Institute for Health and Welfare; Satu Havulinna, PhD, Study Director — Finnish Institute for Health and Welfare; Jaana Lindström, Adjunct prof., Study Director — Finnish Institute for Health and Welfare; Riitta Antikainen, professor, Study Director — Oulu City Health Services; Tiia Ngandu, MD, PhD, Adjunct professor, Study Director — Finnish Institute for Health and Welfare; Tuomo Hänninen, Adjunct prof, Study Director — University of Eastern Finland; Jenni Lehtisalo, PhD, Study Director — Finnish Institute for Health and Welfare; Alina Solomon, MD, PhD, Adjunct professor, Study Director — University of Eastern Finland
Locations (5):
- Finland (5):
  - Finnish Institute for Health and Welfare, Helsinki
  - University of Eastern Finland, Kuopio
  - University of Oulu, Oulu
  - Research Center Mediwest, Seinäjoki
  - Finnish Institute for Health and Welfare, Turku

REFERENCES:
- [Background] Kivipelto M, Ngandu T, Laatikainen T, Winblad B, Soininen H, Tuomilehto J. Risk score for the prediction of dementia risk in 20 years among middle aged people: a longitudinal, population-based study. Lancet Neurol. 2006 Sep;5(9):735-41. doi: 10.1016/S1474-4422(06)70537-3. PMID 16914401
- [Background] Kivipelto M, Helkala EL, Laakso MP, Hanninen T, Hallikainen M, Alhainen K, Soininen H, Tuomilehto J, Nissinen A. Midlife vascular risk factors and Alzheimer's disease in later life: longitudinal, population based study. BMJ. 2001 Jun 16;322(7300):1447-51. doi: 10.1136/bmj.322.7300.1447. PMID 11408299
- [Background] Kivipelto M, Helkala EL, Hanninen T, Laakso MP, Hallikainen M, Alhainen K, Soininen H, Tuomilehto J, Nissinen A. Midlife vascular risk factors and late-life mild cognitive impairment: A population-based study. Neurology. 2001 Jun 26;56(12):1683-9. doi: 10.1212/wnl.56.12.1683. PMID 11425934
- [Background] Kivipelto M, Helkala EL, Laakso MP, Hanninen T, Hallikainen M, Alhainen K, Iivonen S, Mannermaa A, Tuomilehto J, Nissinen A, Soininen H. Apolipoprotein E epsilon4 allele, elevated midlife total cholesterol level, and high midlife systolic blood pressure are independent risk factors for late-life Alzheimer disease. Ann Intern Med. 2002 Aug 6;137(3):149-55. doi: 10.7326/0003-4819-137-3-200208060-00006. PMID 12160362
- [Background] Rovio S, Kareholt I, Helkala EL, Viitanen M, Winblad B, Tuomilehto J, Soininen H, Nissinen A, Kivipelto M. Leisure-time physical activity at midlife and the risk of dementia and Alzheimer's disease. Lancet Neurol. 2005 Nov;4(11):705-11. doi: 10.1016/S1474-4422(05)70198-8. PMID 16239176
- [Background] Kivipelto M, Ngandu T, Fratiglioni L, Viitanen M, Kareholt I, Winblad B, Helkala EL, Tuomilehto J, Soininen H, Nissinen A. Obesity and vascular risk factors at midlife and the risk of dementia and Alzheimer disease. Arch Neurol. 2005 Oct;62(10):1556-60. doi: 10.1001/archneur.62.10.1556. PMID 16216938
- [Background] Lindstrom J, Ilanne-Parikka P, Peltonen M, Aunola S, Eriksson JG, Hemio K, Hamalainen H, Harkonen P, Keinanen-Kiukaanniemi S, Laakso M, Louheranta A, Mannelin M, Paturi M, Sundvall J, Valle TT, Uusitupa M, Tuomilehto J; Finnish Diabetes Prevention Study Group. Sustained reduction in the incidence of type 2 diabetes by lifestyle intervention: follow-up of the Finnish Diabetes Prevention Study. Lancet. 2006 Nov 11;368(9548):1673-9. doi: 10.1016/S0140-6736(06)69701-8. PMID 17098085
- [Background] Kivipelto M, Rovio S, Ngandu T, Kareholt I, Eskelinen M, Winblad B, Hachinski V, Cedazo-Minguez A, Soininen H, Tuomilehto J, Nissinen A. Apolipoprotein E epsilon4 magnifies lifestyle risks for dementia: a population-based study. J Cell Mol Med. 2008 Dec;12(6B):2762-71. doi: 10.1111/j.1582-4934.2008.00296.x. Epub 2008 Feb 8. PMID 18318693
- [Result] Kivipelto M, Solomon A, Ahtiluoto S, Ngandu T, Lehtisalo J, Antikainen R, Backman L, Hanninen T, Jula A, Laatikainen T, Lindstrom J, Mangialasche F, Nissinen A, Paajanen T, Pajala S, Peltonen M, Rauramaa R, Stigsdotter-Neely A, Strandberg T, Tuomilehto J, Soininen H. The Finnish Geriatric Intervention Study to Prevent Cognitive Impairment and Disability (FINGER): study design and progress. Alzheimers Dement. 2013 Nov;9(6):657-65. doi: 10.1016/j.jalz.2012.09.012. Epub 2013 Jan 17. PMID 23332672
- [Result] Ngandu T, Lehtisalo J, Levalahti E, Laatikainen T, Lindstrom J, Peltonen M, Solomon A, Ahtiluoto S, Antikainen R, Hanninen T, Jula A, Mangialasche F, Paajanen T, Pajala S, Rauramaa R, Strandberg T, Tuomilehto J, Soininen H, Kivipelto M. Recruitment and baseline characteristics of participants in the Finnish Geriatric Intervention Study to Prevent Cognitive Impairment and Disability (FINGER)-a randomized controlled lifestyle trial. Int J Environ Res Public Health. 2014 Sep 10;11(9):9345-60. doi: 10.3390/ijerph110909345. PMID 25211775
- [Result] Ngandu T, Lehtisalo J, Solomon A, Levalahti E, Ahtiluoto S, Antikainen R, Backman L, Hanninen T, Jula A, Laatikainen T, Lindstrom J, Mangialasche F, Paajanen T, Pajala S, Peltonen M, Rauramaa R, Stigsdotter-Neely A, Strandberg T, Tuomilehto J, Soininen H, Kivipelto M. A 2 year multidomain intervention of diet, exercise, cognitive training, and vascular risk monitoring versus control to prevent cognitive decline in at-risk elderly people (FINGER): a randomised controlled trial. Lancet. 2015 Jun 6;385(9984):2255-63. doi: 10.1016/S0140-6736(15)60461-5. Epub 2015 Mar 12. PMID 25771249
- [Result] Kulmala J, Ngandu T, Pajala S, Lehtisalo J, Levalahti E, Antikainen R, Laatikainen T, Oksa H, Peltonen M, Rauramaa R, Soininen H, Strandberg T, Tuomilehto J, Kivipelto M. Leisure-Time and Occupational Physical Activity in Early and Late Adulthood in Relation to Later Life Physical Functioning. J Phys Act Health. 2016 Oct;13(10):1079-1087. doi: 10.1123/jpah.2015-0664. Epub 2016 Aug 16. PMID 27254853
- [Result] Strandberg TE, Levälahti E, Ngandu T, Solomon A, M Kivipelto for FINGER Study Group. Health-Related Quality of Life in a Multidomain Intervention Trial to Prevent Cognitive Decline (FINGER). Eur Ger Med. 2017; 8: 164-167.
- [Result] Lehtisalo J, Ngandu T, Valve P, Antikainen R, Laatikainen T, Strandberg T, Soininen H, Tuomilehto J, Kivipelto M, Lindstrom J. Nutrient intake and dietary changes during a 2-year multi-domain lifestyle intervention among older adults: secondary analysis of the Finnish Geriatric Intervention Study to Prevent Cognitive Impairment and Disability (FINGER) randomised controlled trial. Br J Nutr. 2017 Aug;118(4):291-302. doi: 10.1017/S0007114517001982. PMID 28875868
- [Result] Marengoni A, Rizzuto D, Fratiglioni L, Antikainen R, Laatikainen T, Lehtisalo J, Peltonen M, Soininen H, Strandberg T, Tuomilehto J, Kivipelto M, Ngandu T. The Effect of a 2-Year Intervention Consisting of Diet, Physical Exercise, Cognitive Training, and Monitoring of Vascular Risk on Chronic Morbidity-the FINGER Randomized Controlled Trial. J Am Med Dir Assoc. 2018 Apr;19(4):355-360.e1. doi: 10.1016/j.jamda.2017.09.020. Epub 2017 Nov 3. PMID 29108888
- [Result] Solomon A, Handels R, Wimo A, Antikainen R, Laatikainen T, Levalahti E, Peltonen M, Soininen H, Strandberg T, Tuomilehto J, Kivipelto M, Ngandu T. Effect of a Multidomain Lifestyle Intervention on Estimated Dementia Risk. J Alzheimers Dis. 2021;82(4):1461-1466. doi: 10.3233/JAD-210331. PMID 34151805
- [Result] Lehtisalo J, Rusanen M, Solomon A, Antikainen R, Laatikainen T, Peltonen M, Strandberg T, Tuomilehto J, Soininen H, Kivipelto M, Ngandu T. Effect of a multi-domain lifestyle intervention on cardiovascular risk in older people: the FINGER trial. Eur Heart J. 2022 Jun 1;43(21):2054-2061. doi: 10.1093/eurheartj/ehab922. PMID 35051281
- [Result] Wimo A, Handels R, Antikainen R, Eriksdotter M, Jonsson L, Knapp M, Kulmala J, Laatikainen T, Lehtisalo J, Peltonen M, Skoldunger A, Soininen H, Solomon A, Strandberg T, Tuomilehto J, Ngandu T, Kivipelto M. Dementia prevention: The potential long-term cost-effectiveness of the FINGER prevention program. Alzheimers Dement. 2023 Mar;19(3):999-1008. doi: 10.1002/alz.12698. Epub 2022 Jul 16. PMID 35841619
- [Derived] Saaskilahti M, Aarnio E, Levalahti E, Lehtisalo J, Kivipelto M, Strandberg T, Antikainen R, Soininen H, Laatikainen T, Tuomilehto J, Solomon A, Mangialasche F, Ngandu T. Cardiovascular and glucose-lowering medication use among older adults: results from 9-year follow-up of the FINGER trial. Eur Geriatr Med. 2025 Dec 3. doi: 10.1007/s41999-025-01354-1. Online ahead of print. PMID 41339545
- [Derived] Lorenzon G, Marseglia A, Mohanty R, Lehtisalo J, Poulakis K, Ngandu T, Solomon A, Kivipelto M, Westman E. Brain patterns and risk factors in the FINGER RCT multimodal lifestyle intervention. J Prev Alzheimers Dis. 2025 Dec;12(10):100390. doi: 10.1016/j.tjpad.2025.100390. Epub 2025 Sep 24. PMID 40998691
- [Derived] Lorenzo T, Ngandu T, Lehtisalo J, Antikainen R, Gispert JD, Kemppainen N, Laatikainen T, Lindstrom J, Rinne J, Soininen H, Strandberg T, Torre R, Tuomilehto J, Solomon A, Kivipelto M. Associations of Prediabetes, Diabetes and Glucose-Related Markers With Cognition and Neuroimaging in a 2-Year Multidomain Lifestyle Randomised Controlled Trial. Diabetes Metab Res Rev. 2025 Jul;41(5):e70053. doi: 10.1002/dmrr.70053. PMID 40478656
- [Derived] Lehtisalo J, Saaskilahti M, Harkanen T, Kulmala J, Hemio K, Siltanen S, Zhi Z, Mangialasche F, Laatikainen T, Strandberg T, Antikainen R, Tuomilehto J, Soininen H, Kivipelto M, Ngandu T. Changes in older persons' lifestyle and perceived health over time and during the COVID-19 pandemic: findings from the extended follow-up of the FINGER randomized controlled trial from 2009 to 2020. BMC Geriatr. 2025 May 3;25(1):308. doi: 10.1186/s12877-025-05979-6. PMID 40319270
- [Derived] Kekkonen E, Hall A, Antikainen R, Havulinna S, Kivipelto M, Kulmala J, Laatikainen T, Paajanen TI, Sindi S, Soininen H, Strandberg T, Tuomilehto J, Ngandu T, Solomon A. Impaired sleep, depressive symptoms, and pain as determinants of physical activity and exercise intervention adherence: an exploratory analysis of a randomized clinical trial. BMC Geriatr. 2025 Mar 29;25(1):211. doi: 10.1186/s12877-025-05830-y. PMID 40158087
- [Derived] Vaskivuo L, Hokkanen L, Levalahti E, Hanninen T, Antikainen R, Backman L, Laatikainen T, Paajanen T, Stigsdotter Neely A, Strandberg T, Tuomilehto J, Soininen H, Kivipelto M, Ngandu T. Subjective Memory Complaints and the Effect of a Multidomain Lifestyle Intervention on Cognition: The FINGER Trial. J Gerontol B Psychol Sci Soc Sci. 2024 Dec 11;80(1):gbae179. doi: 10.1093/geronb/gbae179. PMID 39450437
- [Derived] Goikolea J, Gerenu G, Daniilidou M, Mangialasche F, Mecocci P, Ngandu T, Rinne J, Solomon A, Kivipelto M, Cedazo-Minguez A, Sandebring-Matton A, Maioli S. Serum Thioredoxin-80 is associated with age, ApoE4, and neuropathological biomarkers in Alzheimer's disease: a potential early sign of AD. Alzheimers Res Ther. 2022 Feb 24;14(1):37. doi: 10.1186/s13195-022-00979-9. PMID 35209952
- [Derived] Alenius M, Ngandu T, Koskinen S, Hallikainen I, Hanninen T, Karrasch M, Kivipelto M, Raivio MM, Laakkonen ML, Kruger J, Suhonen NM, Hokkanen L. Education-Based Cutoffs for Cognitive Screening of Alzheimer's Disease. Dement Geriatr Cogn Disord. 2022;51(1):42-55. doi: 10.1159/000521982. Epub 2022 Feb 23. PMID 35196653
- [Derived] Neuvonen E, Lehtisalo J, Solomon A, Antikainen R, Havulinna S, Hanninen T, Laatikainen T, Lindstrom J, Rautio N, Soininen H, Strandberg T, Tuomilehto J, Kivipelto M, Ngandu T. Psychosocial determinants for adherence to a healthy lifestyle and intervention participation in the FINGER trial: an exploratory analysis of a randomised clinical trial. Aging Clin Exp Res. 2022 Aug;34(8):1793-1805. doi: 10.1007/s40520-022-02088-x. Epub 2022 Feb 19. PMID 35182352
- [Derived] Ngandu T, Lehtisalo J, Korkki S, Solomon A, Coley N, Antikainen R, Backman L, Hanninen T, Lindstrom J, Laatikainen T, Paajanen T, Havulinna S, Peltonen M, Neely AS, Strandberg T, Tuomilehto J, Soininen H, Kivipelto M. The effect of adherence on cognition in a multidomain lifestyle intervention (FINGER). Alzheimers Dement. 2022 Jul;18(7):1325-1334. doi: 10.1002/alz.12492. Epub 2021 Oct 20. PMID 34668644
- [Derived] Sandebring-Matton A, Goikolea J, Bjorkhem I, Paternain L, Kemppainen N, Laatikainen T, Ngandu T, Rinne J, Soininen H, Cedazo-Minguez A, Solomon A, Kivipelto M. 27-Hydroxycholesterol, cognition, and brain imaging markers in the FINGER randomized controlled trial. Alzheimers Res Ther. 2021 Mar 6;13(1):56. doi: 10.1186/s13195-021-00790-y. PMID 33676572
- [Derived] Sindi S, Solomon A, Kareholt I, Hovatta I, Antikainen R, Hanninen T, Levalahti E, Laatikainen T, Lehtisalo J, Lindstrom J, Paajanen T, Peltonen M, Singh Khalsa D, Wolozin B, Strandberg T, Tuomilehto J, Soininen H, Ngandu T, Kivipelto M; FINGER Study Group. Telomere Length Change in a Multidomain Lifestyle Intervention to Prevent Cognitive Decline: A Randomized Clinical Trial. J Gerontol A Biol Sci Med Sci. 2021 Feb 25;76(3):491-498. doi: 10.1093/gerona/glaa279. PMID 33175128
- [Derived] Stephen R, Liu Y, Ngandu T, Antikainen R, Hulkkonen J, Koikkalainen J, Kemppainen N, Lotjonen J, Levalahti E, Parkkola R, Pippola P, Rinne J, Strandberg T, Tuomilehto J, Vanninen R, Kivipelto M, Soininen H, Solomon A; FINGER study group. Brain volumes and cortical thickness on MRI in the Finnish Geriatric Intervention Study to Prevent Cognitive Impairment and Disability (FINGER). Alzheimers Res Ther. 2019 Jun 4;11(1):53. doi: 10.1186/s13195-019-0506-z. PMID 31164160
- [Derived] Kulmala J, Ngandu T, Havulinna S, Levalahti E, Lehtisalo J, Solomon A, Antikainen R, Laatikainen T, Pippola P, Peltonen M, Rauramaa R, Soininen H, Strandberg T, Tuomilehto J, Kivipelto M. The Effect of Multidomain Lifestyle Intervention on Daily Functioning in Older People. J Am Geriatr Soc. 2019 Jun;67(6):1138-1144. doi: 10.1111/jgs.15837. Epub 2019 Feb 26. PMID 30809801
- [Derived] Lehtisalo J, Levalahti E, Lindstrom J, Hanninen T, Paajanen T, Peltonen M, Antikainen R, Laatikainen T, Strandberg T, Soininen H, Tuomilehto J, Kivipelto M, Ngandu T. Dietary changes and cognition over 2 years within a multidomain intervention trial-The Finnish Geriatric Intervention Study to Prevent Cognitive Impairment and Disability (FINGER). Alzheimers Dement. 2019 Mar;15(3):410-417. doi: 10.1016/j.jalz.2018.10.001. Epub 2018 Dec 4. PMID 30527596
- [Derived] Solomon A, Turunen H, Ngandu T, Peltonen M, Levalahti E, Helisalmi S, Antikainen R, Backman L, Hanninen T, Jula A, Laatikainen T, Lehtisalo J, Lindstrom J, Paajanen T, Pajala S, Stigsdotter-Neely A, Strandberg T, Tuomilehto J, Soininen H, Kivipelto M. Effect of the Apolipoprotein E Genotype on Cognitive Change During a Multidomain Lifestyle Intervention: A Subgroup Analysis of a Randomized Clinical Trial. JAMA Neurol. 2018 Apr 1;75(4):462-470. doi: 10.1001/jamaneurol.2017.4365. PMID 29356827